CLINICAL TRIAL: NCT00704184
Title: A Phase II, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of MK7009 Administered Concomitantly With Pegylated-Interferon and Ribavirin for 28 Days in Treatment-Naive Patients With Chronic Hepatitis C Infection
Brief Title: Safety and Efficacy of Vaniprevir (MK7009) Administered With Pegylated-Interferon and Ribavirin (MK-7009-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7009-007; MK7009-007; 2007_658
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Results first posted 2014-10-01 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — vaniprevir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo + Peg-IFN/Ribavirin (Placebo Comparator): Participants took double-blind Placebo + Peg-IFN/Ribavirin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavirin from Week 5 to Week 48.
  Interventions: Drug: Comparator: Pegylated-Interferon (Peg-IFN); Drug: Comparator: Ribavirin
- Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin (Experimental): Participants took double-blind Vaniprevir 300 mg twice daily (b.i.d.) + Peg-IFN/Ribavirin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavirin from Week 5 to Week 48.
  Interventions: Drug: Comparator: Vaniprevir; Drug: Comparator: Pegylated-Interferon (Peg-IFN); Drug: Comparator: Ribavirin
- Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin (Experimental): Participants took double-blind Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavirin from Week 5 to Week 48.
  Interventions: Drug: Comparator: Vaniprevir; Drug: Comparator: Pegylated-Interferon (Peg-IFN); Drug: Comparator: Ribavirin
- Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin (Experimental): Participants took double-blind Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavirin from Week 5 to Week 48.
  Interventions: Drug: Comparator: Vaniprevir; Drug: Comparator: Pegylated-Interferon (Peg-IFN); Drug: Comparator: Ribavirin
- Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin (Experimental): Participants took double-blind Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavirin from Week 5 to Week 48.
  Interventions: Drug: Comparator: Vaniprevir; Drug: Comparator: Pegylated-Interferon (Peg-IFN); Drug: Comparator: Ribavirin; Drug: Comparator: placebo

INTERVENTIONS:
Drug: Comparator: Vaniprevir — Vaniprevir 300 mg b.i.d., 600 mg b.i.d., 600 mg q.d., or 800 mg q.d.; duration of treatment: 28 days
  Other Names: MK-7009
  Arms: Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin; Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin; Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin; Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Drug: Comparator: Pegylated-Interferon (Peg-IFN) — Peg-IFN 180 mcg once-weekly subcutaneous injection; duration of treatment: 48 weeks
Drug: Comparator: Ribavirin — Ribavirin 200 mg tablet b.i.d. (dose based on body weight); duration of treatment: 48 weeks
Drug: Comparator: placebo — Matching placebo to vaniprevir; duration of treatment: 28 days
  Arms: Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin

SUMMARY:
A study to evaluate how effective different levels of Vaniprevir (MK-7009), when administered with Pegylated-Interferon (Peg-IFN) and Ribavirin, are at achieving rapid viral response (RVR) i.e., undetectable hepatitis C virus [HCV] viral ribonucleic acid [RNA] at Week 4 in participants with chronic HCV infection. The primary hypothesis was that the proportion of participants in one or more of the Vaniprevir treatment groups achieving RVR would be greater than the proportion of placebo participants achieving RVR when Vaniprevir and placebo were co-administered with Peg-IFN/Ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Patient has chronic Genotype 1 Hepatitis C infection

Exclusion Criteria:

* Subject has been previously treated for HCV
* Has Human Immunodeficiency Virus (HIV)
* Has Hepatitis B
* Has a history of clinically significant medical condition that may interfere with the study (e.g., stroke or chronic seizures or major neurological disorder) or is contraindicated for treatment with peg-IFN and Ribavirin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-07-25 (Actual); Primary Completion 2008-12-12 (Actual); Study Completion 2010-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Manns MP, Gane E, Rodriguez-Torres M, Stoehr A, Yeh CT, Marcellin P, Wiedmann RT, Hwang PM, Caro L, Barnard RJ, Lee AW; MK-7009 Protocol 007 Study Group. Vaniprevir with pegylated interferon alpha-2a and ribavirin in treatment-naive patients with chronic hepatitis C: a randomized phase II study. Hepatology. 2012 Sep;56(3):884-93. doi: 10.1002/hep.25743. Epub 2012 Jul 17. PMID 22473713
- [Derived] Lawitz E, Sulkowski M, Jacobson I, Kraft WK, Maliakkal B, Al-Ibrahim M, Gordon SC, Kwo P, Rockstroh JK, Panorchan P, Miller M, Caro L, Barnard R, Hwang PM, Gress J, Quirk E, Mobashery N. Characterization of vaniprevir, a hepatitis C virus NS3/4A protease inhibitor, in patients with HCV genotype 1 infection: safety, antiviral activity, resistance, and pharmacokinetics. Antiviral Res. 2013 Sep;99(3):214-20. doi: 10.1016/j.antiviral.2013.05.015. Epub 2013 Jun 7. PMID 23747481
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=7009-007&kw=7009-007&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the double-blind phase (Day 1 to Day 28), participants took Vaniprevir or Placebo in combination with Pegylated Interferon (Peg-IFN)/Ribavirin. During the open-label phase (Day 29 to Week 48), participants took Peg-IFN/Ribavirin only.
Groups:
- Placebo + Peg-IFN/Ribavirin: Participants took double-blind Placebo + Peg-IFN/Ribavarin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavarin from Week 5 to Week 48.
- Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin: Participants took double-blind Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavarin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavarin from Week 5 to Week 48.
- Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin: Participants took double-blind Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavarin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavarin from Week 5 to Week 48.
- Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin: Participants took double-blind Vaniprevir 600 mg q.d. + Peg-IFN/Ribavarin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavarin from Week 5 to Week 48.
- Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin: Participants took double-blind Vaniprevir 800 mg q.d. + Peg-IFN/Ribavarin from Week 1 to Week 4, followed by open-label Peg-IFN/Ribavarin from Week 5 to Week 48.
Period: Double-Blind Treatment
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Started | 20 | 18 | 20 | 18 | 19
Treated | 19 (One participant was randomized to placebo but withdrew prior to receiving study medication.) | 18 | 20 | 18 | 19
Completed | 19 | 18 | 20 | 18 | 19
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Period: Open-Label Treatment
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Started | 19 | 18 | 20 | 18 | 19
Completed | 18 | 16 | 16 | 13 | 16
Not Completed | 1 | 2 | 4 | 5 | 3
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 2 | 2 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population consists of all participants treated with study medication. One participant was randomized to the placebo group but withdrew from the study prior to taking any study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin | Total
Number analyzed (Participants) | 19 | 18 | 20 | 18 | 19 | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.8 (10.1) | 46.7 (10.2) | 42.0 (10.7) | 50.1 (8.4) | 45.1 (12.0) | 46.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 9 | 11 | 7 | 39
  Male | 11 | 14 | 11 | 7 | 12 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving RVR
Description: Rapid Viral Response (RVR) was declared if Hepatitis C Virus (HCV) ribonucleic acid (RNA) was undetectable at Week 4.
Time Frame: Week 4
Population: The Per Protocol population included all participants who did not have clinically important deviations from protocol-specified criteria. Only participants with an HCV RNA result at the Week 4 time point were included in the analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Number analyzed (Participants) | 18 | 16 | 19 | 16 | 18
Percentage of Participants | 5.6 | 75.0 | 78.9 | 68.8 | 83.3
Statistical Analysis 1: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted difference in % = 69.3, 95% CI 2-sided [40.3 to 86.7] — Adjusted difference subtracts the percentage of placebo responders (5.3%) and stratifies by HCV genotype (1a vs. non-1a)
Statistical Analysis 2: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted difference in % = 73.6, 95% CI 2-sided [46.0 to 88.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted difference in % = 63.3, 95% CI 2-sided [32.8 to 82.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; p < 0.001, Miettinen and Nurminen method; Adjusted difference in % = 77.8, 95% CI 2-sided [49.2 to 91.3] — Adjusted difference subtracts the percentage of placebo responders (5.3) and stratifies by HCV genotype (1a vs. non-1a)

2. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: The number of participants experiencing AEs in each treatment group was monitored during the Vaniprevir/Placebo treatment (Day 1 to Day 28) and safety follow-up (Day 29 to Day 42) periods.
Time Frame: Up to Day 42
Population: The Safety Population consists of all randomized participants who received at least 1 dose of study therapy.
Measure: Number; unit: Participants
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Number analyzed (Participants) | 19 | 18 | 20 | 18 | 19
Participants | 18 | 15 | 18 | 16 | 18

3. Primary Outcome: Number of Participants Discontinuing From Study Therapy Due to AEs
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of study therapy, whether or not considered related to the use of the product.
Time Frame: Day 1 to Day 28
Population: The Safety Population consists of all randomized participants who received at least 1 dose of study therapy
Measure: Number; unit: Participants
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Number analyzed (Participants) | 19 | 18 | 20 | 18 | 19
Participants | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With ≥2-log10 Decrease in HCV RNA
Description: The number of participants with at least a 2-log10 decrease from baseline in HCV RNA following 4 weeks of treatment with Placebo or Vaniprevir.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Number analyzed (Participants) | 18 | 16 | 19 | 16 | 18
Number of Participants | 16 | 16 | 19 | 16 | 17
Statistical Analysis 1: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Adjusted difference = 11.2, 95% CI 2-sided [-9.7 to 33.8] — Adjusted difference subtracts the percentage of placebo responders (88.9%) and stratifies by HCV genotype (1a vs. non-1a)
Statistical Analysis 2: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Adjusted difference = 10.8, 95% CI 2-sided [-7.6 to 33.2] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Adjusted difference = 11.2, 95% CI 2-sided [-9.7 to 33.8] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Adjusted difference = 5.4, 95% CI 2-sided [-16.5 to 28.4] — [estimate comment as in outcome 4, analysis 1]

5. Secondary Outcome: Number of Participants With ≥3-log10 Decrease in HCV RNA
Description: The number of participants with at least a 3-log10 decrease from baseline in HCV RNA following 4 weeks of treatment with Placebo or Vaniprevir.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Number analyzed (Participants) | 18 | 16 | 19 | 16 | 18
Number of Participants | 15 | 16 | 19 | 16 | 17
Statistical Analysis 1: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Adjusted difference = 16.9, 95% CI 2-sided [-4.0 to 40.2] — Adjusted difference subtracts the percentage of placebo responders (83.3%) and stratifies by HCV genotype (1a vs. non-1a)
Statistical Analysis 2: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Adjusted difference = 16.2, 95% CI 2-sided [-2.2 to 39.5] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Adjusted difference = 16.9, 95% CI 2-sided [-4.0 to 40.2] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Adjusted difference = 10.7, 95% CI 2-sided [-11.4 to 34.6] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Mean Log Change From Baseline in HCV RNA
Description: The mean changes from baseline in log10 HCV RNA in each vaniprevir group was compared against control treatment at Week 4.
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Number analyzed (Participants) | 18 | 16 | 19 | 17 | 18
Log10 IU/mL | -3.6 (1.3) | -6.1 (1.1) | -6.3 (0.7) | -6.2 (0.6) | -6.3 (1.4)
Statistical Analysis 1: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Difference in Least Squares (LC) Means = -2.5, 95% CI 2-sided [-3.2 to -1.8] — The difference in LS Means reflects the mean decrease from baseline in HCV RNA between vaniprevir and placebo at Week 4
Statistical Analysis 2: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Difference in LS Means = -2.7, 95% CI 2-sided [-3.4 to -2.0] — The difference in LS Means reflects the mean decrease from baseline in HCV RNA between vaniprevir and placebo at Week 4
Statistical Analysis 3: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Difference in LS Means = -2.7, 95% CI 2-sided [-3.4 to -2.0] — The difference in LS Means reflects the mean decrease from baseline in HCV RNA between vaniprevir and placebo at Week 4
Statistical Analysis 4: Comparison: Placebo + Peg-IFN/Ribavirin vs Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin; Test type: Superiority or Other; Difference in LS Means = -2.7, 95% CI 2-sided [-3.3 to -2.0] — The difference in LS Means reflects the mean decrease from baseline in HCV RNA between vaniprevir and placebo at Week 4

ADVERSE EVENTS:
Time Frame: AEs were monitored for 18 months in the study, including the Vaniprevir/Placebo + Peg-IFN Ribavirin treatment/follow-up period (Day 1 to Day 42) and subsequent Peg-IFN/Ribavirin treatment/follow-up period (Day 43 to Week 72).
Description: The Safety Population consists of all randomized participants who received at least 1 dose of study therapy.
Arm/Group | Placebo + Peg-IFN/Ribavirin | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin
Serious Adverse Events (participants affected / at risk) | 1/19 | 3/18 | 1/20 | 2/18 | 2/19
Other Adverse Events (participants affected / at risk) | 19/19 | 16/18 | 20/20 | 17/18 | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Peg-IFN/Ribavirin (N=19) | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin (N=18) | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin (N=20) | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin (N=18) | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin (N=19)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Peg-IFN/Ribavirin (N=19) | Vaniprevir 300 mg b.i.d. + Peg-IFN/Ribavirin (N=18) | Vaniprevir 600 mg b.i.d. + Peg-IFN/Ribavirin (N=20) | Vaniprevir 600 mg q.d. + Peg-IFN/Ribavirin (N=18) | Vaniprevir 800 mg q.d. + Peg-IFN/Ribavirin (N=19)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vision acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual brightness (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Xerophthalmia (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 2 (2) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 1 (1) | 3 (3) | 4 (4) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 7 (8) | 2 (2) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 4 (4) | 0 (0) | 2 (2) | 4 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrooesophogeal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip erosion (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 5 (7) | 8 (14) | 7 (8) | 6 (6)
Oesophogeal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 9 (16) | 4 (5) | 3 (6)
Asthenia (General disorders) | 4 (5) | 2 (2) | 4 (6) | 4 (4) | 3 (3)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Chills (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 7 (7) | 3 (3) | 7 (10) | 4 (4) | 3 (3)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 4 (5) | 4 (4) | 4 (4) | 4 (4) | 5 (6)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Injection site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 3 (4) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Mucosal dryness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (5)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Glucose urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 4 (4) | 6 (6) | 2 (2) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 2 (4) | 3 (3) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (10) | 4 (4) | 9 (12) | 8 (9) | 5 (6)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysthymic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4) | 4 (4) | 5 (5) | 2 (2)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4) | 2 (3) | 2 (2) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 1 (2)
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Hypotrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (8) | 4 (4) | 0 (0) | 1 (1) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (6) | 2 (2) | 3 (3) | 2 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular icterus (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication guidelines.